CLINICAL TRIAL: NCT00472004
Title: A Prospective, Randomized, Open Label Study To Compare The Efficacy, Safety And Tolerability Of 17-B Estradiol/Trimegestone CC 1 Mg (Totelle) And Tibolone (Livial) In Postmenopausal Women.
Brief Title: Study Comparing 17B Estradiol/TMG CC 1mg Vs. Tibolone In Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0753T-101800; B2481004
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Vasomotor Symptoms
MeSH Terms: interventions — tibolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 17B Estradiol (1mg) / (0.125 mg) Trimegestone (TMG) Continuous combined, 1 Daily, 1 year duration
  Interventions: Drug: 17B Estradiol (1mg) / (0.125 mg) TMG Continuous combined (Totelle)
- 2 (Active Comparator): Tibolone 2.5 mg 1 daily, 1 year duration
  Interventions: Drug: Tibolone (Livial)

INTERVENTIONS:
Drug: 17B Estradiol (1mg) / (0.125 mg) TMG Continuous combined (Totelle) — 17B Estradiol (1mg) / (0.125 mg) TMG Continuous combined, 1 Daily, 1 year duration
  Other Names: Totelle
  Arms: 1
Drug: Tibolone (Livial) — Tibolone 2.5 mg 1 daily, 1 year duration
  Other Names: Livial
  Arms: 2

SUMMARY:
This is a Phase IV prospective, randomized, open label, comparative, multicenter study in generally healthy postmenopausal women receiving Totelle (17B Estradiol/TMG CC (1mg)) and Livial (Tibolone).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy postmenopausal women
* Last natural (without exogenous hormone therapy) menstrual cycle completed at least 12 consecutive months prior to screening and without any other kind of gynecological bleeding during this same period
* At least 1 year of natural occurring amenorrhea

Exclusion Criteria:

* Known or suspected estrogen-dependent neoplasia
* Endometrial hyperplasia
* Any malignancy with the exception of a history of basal cell carcinoma of the skin

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Decreased of Vasomotor Symptoms [from baseline to six and twelve months] | 1 year

SECONDARY OUTCOMES:
Changes in Body Weight (from baseline to six and twelve months) | 1 year
Quality of Life (from baseline to six and twelve months) | 1 year
Treatment Adherence (from baseline to six and twelve months) | 1 year
Breast Tenderness (from baseline to six and twelve months) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0753T-101800&StudyName=Study%20Comparing%2017B%20Estradiol/TMG%20CC%201mg%20Vs.%20Tibolone%20In%20Postmenopausal%20Women